CLINICAL TRIAL: NCT02463019
Title: An Open-label Rollover Study in Chinese Patients After Finishing a 3-year Randomize Trial for Chronic Hepatitis B With High Serum Viral Load But Mild Elevated Aminotransferase
Brief Title: Roll-over After 3-year Trial for Tenofovir in Mild Chronic Hepatitis B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: E-DA Hospital (Other)
Collaborators: Taipei Institute of Pathology (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDAHospital
Record Dates: First submitted 2015-05-14; First posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Hepatitis B; Antiviral Treatment
Keywords: hepatitis B virus; tenofovir
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tenofovir (Other): Tenofovir Disoproxil Fumarate 300mg daily for 3 years
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Tenofovir Disoproxil Fumarate
  Other Names: Viread

SUMMARY:
This open-label study is an roll-over extension of a randomized trial "Efficacy of Tenofovir Disoproxil Fumarate in Chronic Hepatitis B Patients with High Viral Load but Slight Aminotransferase Elevation" (NCT01522625).

After finishing the 3-year therapeutic trial, all patients receive open-label TDF for another 3 years. All patients undergo liver biopsy to evaluate the stage of fibrosis after the 3-year open-label therapy. During the 3-year period, patients were followed up every 12 weeks for the biochemical, serological, virological parameters, and adverse reactions.

The primary outcome is the progression of liver fibrosis. Safety issues such as change of renal function and bone mineral density are 2nd outcomes.

DETAILED DESCRIPTION:
Background The indication to start NUCs remains controversial in non-cirrhotic compensated patients with chronic hepatitis B (CHB). Specifically, it has not been clarified whether high serum concentration of HBV DNA warrants treatment despite only mild elevation of serum alanine aminotransferase (ALT). In order to elucidate this unresolved issue, we've conducted a double blind placebo controlled randomized trial to investigate the efficacy of Tenofovir Disoproxil Fumarate (TDF) in CHB patients with high viral load but only mildly elevated serum ALT.

This open-label rollover study is an extension of the aforementioned randomized trial. For those who are initially randomized to placebo and later receive open-label TDF, there is a rare opportunity to study the efficacy of TDF by using the same patient as his/her own control. For those already randomized to TDF in the trial, the investigators will be able to closely monitor all aspects of therapeutic responses (i.e., biochemical, virological, serological, and histological) during a 6-year treatment course in an Asian cohort.

Regardless of their initial treatment assignment, these enrolled patients offer a unique opportunity to further explore the effectiveness of TDF in CHB in that they have paired biopsied liver tissue and comprehensive information.

Objectives:

The primary endpoint of this study is the evolution of liver fibrosis during the therapeutic course. The secondary endpoints are virological response including not only serum viral load but also intracellular HBV markers such as viral covalently closed circular (ccc) DNA, serological response including HBsAg seroconversion, HBeAg seroconversion, and quantification of HBsAg, biochemical response such as AST, ALT, and adverse reactions with particular attention to clinical events regarding bone and renal safety.

Occurrence of drug resistance is also an important end point.

Methods:

After enrollment, all patients are interviewed with a structured questionnaire to obtain information regarding demographic data, social-economic status, life style, and medical history. Physical checkup, hemogram, blood biochemistry, serology of HBV, serum viral load, HBV genotype, and abdominal sonography are performed at baseline.

Enrolled patients are followed up by telephone or interview every 4 weeks and physically examined every 12 weeks. At each follow-up visit, patients are instructed to return the untaken drugs. A patient is defined as compliant if she or he completes at least 80% of the drugs. AST, ALT, HBV DNA, and quantitative HBsAg will be measured every 12 weeks. Serum biochemistry (bilirubin, PT, P, K, Cre), urinalysis, alpha-fetoprotein, HBeAg, and anti-HBe and abdominal sonography are measured every 24 weeks. Hemogram and anti-HBs will be checked annually.

Percutaneous liver biopsy will be performed at the beginning of this project and after completing the 3-year (156 weeks) trial period. Serology of HBV (HBsAg, anti-HBs, HBeAg, and anti-HBe) is determined by commercially available immunoassays (ABBOTT GmbH& Co., Wiesbaden, Germany). Serum HBV DNA is measured quantitatively by quantitative polymerase chain reaction method (Roche COBAS TaqMan Assay). Histopathological specimens obtained by liver biopsy will be evaluated independently by two central histopathologists who are unaware of patients' clinical information. The final report of liver histology is based on the agreement of these two pathologists and if necessary a third pathologist may be invited to settle disagreement.

Analysis Both Intent-to-treat (ITT) and per-protocol (PP) analyses will be performed to assess therapeutic efficacy. All randomized patients are included in the ITT analysis and all protocol violators (compliance less than 80%, loss to follow-up, withdrawal from study) will be excluded from PP analysis. Quantitative data are summarized as mean ± standard deviation (SD) and categorical variables as percentages. Fisher's exact test is used to compare proportions of categorical variables. Unpaired and paired student's t-tests are used to compare means of continuous variables between groups and within groups respectively.

The investigators will apply a multiple logistic regression analysis to investigate factors associated with therapeutic efficacy. All tests are two-tailed and a p value less than 0.05 is considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* all participants should have finished the clinical trial <Efficacy of Tenofovir Disoproxil Fumarate in Chronic Hepatitis B Patients with High Viral Load but Slight Aminotransferase Elevation> without drop-out.
* willingness to adhere to treatment and follow-up plans

Exclusion Criteria:

* co-infection with HIV, HCV, or HDV
* presence of cirrhosis on histopathology
* hepatic decompensation defined as serum bilirubin > 2mg/dl and prolonged prothrombin time > 3 seconds
* concurrent malignant diseases including hepatocellular carcinoma
* severe co-morbidity with life expectancy < 1year
* pregnant or lactating women
* organ transplantation except cornea or hair transplant
* suspected or confirmed chronic liver diseases from etiologies other than HBV (e.g. alcoholic hepatitis, Wilson disease, Hemochromatosis…etc)
* serum creatinine >1.5mg/dL
* refusal to undergo liver biopsy
* lack of informed consent

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change of liver histopathology | 3 years
  evaluated by Knodell and Ishak scoring system

SECONDARY OUTCOMES:
Virological response | 3 years
  HBV DNA undetectability
Drug resistance | 3 years
  elevation of serum viral DNA > 10 folds above nadir during therapy and signature mutation confirmed by viral genetic assay

CONTACTS AND LOCATIONS:
Overall Officials: Jaw-Town Lin, MD., PhD, Study Chair — Fu Jen Catholic University

REFERENCES:
- [Derived] Hsu YC, Chen CY, Tseng CH, Chen CC, Lee TY, Bair MJ, Chen JJ, Huang YT, Chang IW, Chang CY, Wu CY, Wu MS, Mo LR, Lin JT. Antiviral therapy for chronic hepatitis B with mildly elevated aminotransferase: A rollover study from the TORCH-B trial. Clin Mol Hepatol. 2025 Jan;31(1):213-226. doi: 10.3350/cmh.2024.0640. Epub 2024 Oct 17. PMID 39415599